CLINICAL TRIAL: NCT06202040
Title: The Effect of Bilateral Rectus Sheath and Oblique Subcostal Transversus Abdominis Plane Block on Mechanical Power in Patients Undergoing Laparoscopic Cholecystectomy Surgery
Brief Title: The Effect of Bilateral Rectus Sheath and Oblique Subcostal Transversus Abdominis Plane Block on Mechanical Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Esma Karaarslan, Medical Doctor, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MacPower
Record Dates: First submitted 2023-12-21; First posted 2024-01-11 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Mechanical Power

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1:OSTAPand RSB (Active Comparator): Group 1 will consist of patients who received general anesthesia, and just before the surgery started, bilateral OSTAP and RSB will be performed.
  Interventions: Procedure: Bilateral Oblique Subcostal Transversus Abdominis Plane Block (OSTAP) will be performed.; Procedure: Bilateral Rectus Sheath Block (RSB) will be performed.
- Group 2: Intravenous analgesia (No Intervention): Group 2 will include patients who received general anesthesia and were administered intravenous analgesia approximately 30 minutes before the end of the operation.

INTERVENTIONS:
Procedure: Bilateral Oblique Subcostal Transversus Abdominis Plane Block (OSTAP) will be performed. — The OSTAP block will be conducted in-plane using a 100mm 22 G needle and a linear probe under ultrasound (USG) guidance. The 20cc block will contain 10cc of 0.5% bupivacaine and 10cc of normal saline. Bilateral OSTAP will be administered with 20cc (10cc per side). To apply the block, position the linear probe parallel to the rib edge immediately below it on the anterior abdominal wall. Visible will be the external, internal, transversus abdominis, and rectus muscle junction. The needle tip will move toward the TAP space (between the internal oblique and transversus abdominis muscles). To ensure medication delivery, the needle tip will be visible in the TAP and the drug will be aspirated negatively. USG will also observe drug distribution at the rectus abdominis muscle-TAP space junction.
  Arms: Group 1:OSTAPand RSB
Procedure: Bilateral Rectus Sheath Block (RSB) will be performed. — When the patient is in the supine position, the ultrasound (USG) linear probe is held in the transverse plane at the level just above the umbilicus, where the posterior rectus sheath is best visualized. Using the in-plane technique with a 100mm 22 G needle under USG guidance, the drug prepared will be administered between the rectus muscle and the posterior rectus sheath. For this block, a volume of 20cc will be prepared, consisting of 10cc of 0.5% bupivacaine and 10cc of normal saline. Bilateral Rectus Sheath Block (RSB) will be applied with a total volume of 20cc, 10cc to each side.
  Arms: Group 1:OSTAPand RSB

SUMMARY:
The respiratory system receives mechanical power (MP) throughout time during mechanical ventilation. Despite its life-saving benefits, mechanical ventilation can cause ventilator-induced lung injury (VILI). Recently, VILI has been linked to mechanical power, or the amount of energy the mechanical ventilator sends to the respiratory system in a given time. The hunt for lung damage-reducing characteristics, notably after VILI and ARDS (Acute respiratory distress syndrome), has increased after Covid-19. Mechanical power must be used more to promote lung protection. We examined the effects of bilateral rectus sheath and OSTAP (Oblique Subcostal Transversus Abdominis Plane ) block on mechanically powered patients.

DETAILED DESCRIPTION:
MP is the energy transmitted over time to the respiratory system during mechanical ventilation. Although mechanical ventilation is a life-supporting treatment, it has the potential to cause damage to the lung structure in a process referred to as VILI. Recently, the degree of VILI has been associated with the amount of energy transmitted to the respiratory system by the mechanical ventilator within a specific time frame, which is referred to as mechanical power. After the occurrence of Covid-19, the search for parameters to reduce lung damage, especially following VILI and ARDS, has become more prominent. In this regard, promoting lung protection requires the more widespread use of mechanical power. We aimed to investigate the effect of bilateral rectus sheath and OSTAP block applied to patients on mechanical power.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years
* ASA 1-2 patients
* Patients undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* Mental retardation,
* Severe presence of COPD,
* Uncontrolled Bronchial Asthma,
* Decompensated Heart Failure (NYHA 3-4),
* History of previous lung surgery,
* Patients unwilling to participate in the study,
* Local anesthetic allergy,
* History of chronic pain and treatment,
* Morbid obesity (body mass index (BMI) >35),
* Pregnancy,
* Patients converted to open cholecystectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
mechanical power will be calculated from these measurements (mec power 1, mec power 2, mec power 3) as a joule. | Comen after intubation (before the block procedure), end of the surgery pre sugammadex administration and end of the surgery post sugammadex administration
  Primary outcome measures will be based on intraoperative measurements taken from the mechanical ventilator, and mechanical power will be calculated from these measurements (mec power 1, mec power 2, mec power 3).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for pain evaluation (0-10, 0 = no pain, 10 = the most severe pain). | postoperative assessments at 30 minutes, 2 hours, 8 hours, and 24 hours
  Secondary outcome measures will include postoperative assessments at 30 minutes, 2 hours, 8 hours, and 24 hours, using the Visual Analog Scale (VAS) for pain evaluation (0-10, 0 = no pain, 10 = the most severe pain).
the Quality of Recovery-15 Test (QoR-15T) [ Excellent (QoR-15 > 135 point), Good (122 ≤ QoR-15 ≤ 135 points), Moderate (90 ≤ QoR-15 ≤ 121 point), Poor (QoR-15 < 90 points) ] | Postoperative assessments at 24 hours
  Secondary outcome measures will include postoperative assessments at 24 hours, the Quality of Recovery-15 Test (QoR-15T) will be used to assess patient recovery quality.
Number of rescue analgesic needs | Postoperative assessments at 30 minutes, 2 hours, 8 hours, and 24 hours
  Secondary outcome measures will include postoperative assessments at 30 minutes, 2 hours, 8 hours, and 24 hours, number of rescue analgesic needs will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Esma Karaarslan, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya Cıty Hospıtal, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Maybe, we can share all info after finish the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We want to descrıbe time frame after finish the study.
Access Criteria: We can share the data by usın e-mail.

REFERENCES:
- [Derived] Karaarslan E, Tire Y, Tutar MS, Akinci N, Mermer HA, Uyar S, Ates D, Simsek G, Kozanhan B. The effect of bilateral rectus sheath and oblique subcostal transversus abdominis plane blocks on mechanical power in patients undergoing laparoscopic cholecystectomy surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Apr 16;25(1):186. doi: 10.1186/s12871-025-03062-6. PMID 40241019